CLINICAL TRIAL: NCT06357117
Title: Pattern and Extent of Intrahepatic Infiltration of Perihilar Cholangiocarcinoma - A Liver Panoramic Digital Pathological Study
Brief Title: Extent of Intrahepatic Infiltration of Perihilar Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Shuo Jin, Attending physician, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: A01263
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Perihilar Cholangiocarcinoma
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No RLI vs RLI: No RLI: PHCC patients without RLI. RLI: PHCC patients with RLI.
- No DIHI vs DIHI: No DIHI: PHCC patients without DIHI. DIHI: PHCC patients with DIHI.

SUMMARY:
The extent of intrahepatic infiltration of perihilar cholangiocarcinoma (PHCC) remains unclear. This research aimed to explore the pattern and extent of intrahepatic infiltration of PHCC to guide surgical treatment and pathological research. This prospective study included 62 participants diagnosed with PHCC who underwent major hepatectomy. A whole-mount digital liver pathology system (WDLPS) for hepatectomy specimens greater than 10 × 10 cm was used to panoramically assess the intrahepatic infiltration extent of PHCC.

DETAILED DESCRIPTION:
Perihilar cholangiocarcinoma (PHCC) is the most common type of bile duct malignancy, and radical surgical resection is the most effective treatment. The extent and characteristics of the intrahepatic infiltration of PHCC remain unclear, leading to controversy about the extent of liver resection for PHCC. The expert consensus statement of PHCC recommends tumor-invaded lobectomy as the standard procedure for liver resection, however, many studies recommend major hepatectomy (hemihepatectomy or trisectionectomy). Recently, minor hepatectomy has emerged for PHCC, such as resection of segment IVB+V and perihilar combined with segment I resection; however, the efficacy remains controversial. To determine the extent and characteristics of intrahepatic infiltration of PHCC, the investigators constructed a whole-mount digital liver pathology system (WDLPS) that allows the tumor and surrounding liver tissue from major hepatectomy specimens to be displayed in one large section, which could localize the margin of the main tumor and observe the distribution of adenocarcinoma panoramically. In addition, digital measurement was used to accurately measure the range of intrahepatic infiltration to guide the scope of hepatectomy. From April 2018 to December 2021, 62 participants were diagnosed for PHCC based on clinical manifestations, imaging, and pathological findings. All participants underwent hemihepatectomy or trisectionectomy combined with caudate lobectomy. Skeletonization resection of the hepatoduodenal ligament, including dissection of the regional lymph nodes, was performed from the duodenum to the liver. Clinical and pathological indicators of the participants were collected. Portal vein and hepatic artery invasion were defined as the primary or secondary branch in the resected side or the reserved side which was invaded. In this study, the investigators established a WDLPS to study the intrahepatic invasion range and pathway of PHCC through the major hepatectomy specimens panoramically. The distal intrahepatic infiltration (DIHI) and radial liver invasion (RLI) were important components of intrahepatic infiltration of PHCC explored by WDLPS. RLI distance was defined as the maximum straight-line distance from the infiltrated liver parenchyma to the hepatic hilar plate. DIHI was defined as the intrahepatic infiltration greater than 1 cm from the margin of the main tumor. The distance between the DIHI and the margin of the main tumor was recorded. Categorical variables are expressed as percentages (%) and the difference were tested using the chi-squared test or Fisher's exact test. Continuous variables are presented in the form of mean±standard deviation and were tested using the t-test or Mann-Whitney U test, when appropriate. Relapse-free survival (RFS) and Overall survival (OS) were estimated using the Kaplan-Meier method, and differences between groups were assessed by the log-rank test. In addition, the investigators estimated restricted mean survival time (RMST) without a truncation time and RMST differences (ΔRMSTs) for RFS and OS between treatment groups to provide clinically relevant intuitive estimation. Statistical analyses were performed using the SPSS software (version 26.0, SPSS Inc., IBM, Armonk, NY, USA) and R (version 4.2.2.R Core Team.2022).

ELIGIBILITY:
Inclusion Criteria:

1. Patients were diagnosed for PHCC based on clinical manifestations, imaging, and pathological findings.
2. Hepatectomy was performed.
3. WDLPS was successfully produced.

Exclusion Criteria:

1. Not PHCC patients.
2. Patients with PHCC did not undergo hepatectomy.
3. WDLPS was not successfully produced.

Ages: 44 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed for PHCC based on clinical manifestations, imaging, and pathological findings. All patients underwent hemihepatectomy or trisectionectomy combined with caudate lobectomy. Skeletonization resection of the hepatoduodenal ligament, including dissection of the regional lymph nodes, was performed from the duodenum to the liver. Clinical and pathological indicators of the patients were collected. Portal vein and hepatic artery invasion were defined as the primary or secondary branch in the resected side or the reserved side which was invaded.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival (RFS). | RFS as of December 2023
  Refers to the survival time of a PHCC patient without recurrence of PHCC for a period of time after surgical treatment.

SECONDARY OUTCOMES:
Overall survival (OS). | OS as of December 2023
  Refers to the time from the start of surgical treatment to death or the last follow-up of a PHCC patient.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Jin, PhD, Principal Investigator — Beijing Tsinghua Changgung Hospital affiliated to Tsinghua University
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Jin S, Jiang N, Zhao JM, Xiao Y, Wang SY, Xiang CH, Lu Q, Shan SQ, Ruan HT, Yu SQ, Zeng JP, Yang SZ, Li L, Dong JH. Pattern and extent of intrahepatic infiltration of perihilar cholangiocarcinoma - a case-control study based on liver panoramic digital pathology. Int J Surg. 2025 Jan 1;111(1):31-39. doi: 10.1097/JS9.0000000000002040. PMID 39166939